CLINICAL TRIAL: NCT00001440
Title: Pilot Study of Autologous T Cells and/or IL-2 for the Enhancement of Immune Reconstitution After Dose-Intensive Chemotherapy for Breast Cancer
Brief Title: Autologous T-Cell Transplantation and the Immunotherapy of Residual Disease in Breast Cancer: Pilot Study of Vaccine-Driven T-Cell Expansion in Patients Treated With Dose-Intensive Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 950146; 95-C-0146
Record Dates: First submitted 2006-07-13; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-01

CONDITIONS: Breast Neoplasm; Neoplasm Metastasis
Keywords: p53; Interleukin-2; T-Cell Repopulation; Apheresis; RAS
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Interleukin-2

INTERVENTIONS:
Procedure: Autologous T cells
Drug: Interleukin-2

SUMMARY:
The ability of chemotherapy to cure cancer, including breast cancer, has been limited by drug resistant residual tumor cells remaining after chemotherapy that generally result in relapse. Additional therapeutic strategies to eradicate these residual tumor cells are needed. The augmentation of specific anti-tumor immune responses, such as those mediated by T-cells, might represent such an additional strategy for the control or elimination of residual tumor cells. This approach might be especially effective if T-cell mediated responses were enhanced during both the period of T-cell repopulation that follows acute T-cell depletion and in the setting of minimal residual tumor burden present after dose intensive chemotherapy. Such chemotherapy is known to result in severe T-cell depletion. This pilot study has been designed to examine the feasibility of combining dose intensive chemotherapy with interventions aimed at the reconstitution of T-cell immunity. Metastatic or adjuvant breast cancer patients who have received dose intensive chemotherapy will subsequently receive a combination of autologous chemotherapy-naive T-cells, a patient-specific tumor antigen vaccine, and recombinant human interleukin-2. These interventions will be assessed for their ability to modulate T-cell number, T-cell function, and T-cell specificity during the period of T-cell repopulation. Such modulation may result in the effective reconstitution of generalized T-cell immunity with the generation of vaccine-specific anti-tumor T-cell responses.

DETAILED DESCRIPTION:
The process of T cell immune reconstitution post-chemotherapy in breast cancer patients is impaired. Such a deficit in T cell immunity likely represents an important obstacle to tumor vaccine therapy in breast cancer patients. In an attempt to enhance T cell immune reconstitution, we have administered cryopreserved T cells and interleukin-2 to breast cancer patients post-chemotherapy. Initial data from the first 13 patients enrolled on this study suggests that the administration of T cells and IL-2 resulted in improved T cell reconstitution relative to untreated patients or patients receiving only IL-2. Importantly, recipients of the combination of T cells and IL-2 had an enhanced recovery of CD4+CD45RA+ T cells; because this T cell subset represents a naive T cell phenotype that generally maintains a capacity to respond to antigen, enhanced regeneration of this population may result in improved immune function and may allow for a more successful immune response to tumor vaccines. It will be important to now evaluate what effect T cell administration alone (without IL-2 treatment) has on immune reconstitution post-chemotherapy. Determination of the relative benefits of T cell and/or cytokine administration on T cell recovery post-chemotherapy may assist in the development of breast cancer vaccine protocols where a T cell-mediated immune response may be necessary for optimal response to the vaccine.

ELIGIBILITY:
PRE-CHEMOTHERAPY ELIGIBILITY:

Patients must have a histologically confirmed diagnosis of stage II, III, or IV infiltrating breast cancer; stage II patients must be considered high risk with greater than four positive axillary lymph nodes at primary surgery. Patients with metastatic disease must have their relapse confirmed pathologically. All pathological material must be reviewed and the diagnosis confirmed by the Department of Pathology at the NIH Clinical Center prior to acceptance on the protocol.

Patients enrolled on this protocol may receive chemotherapy by one of the following mechanisms: (1) Any dose intensive chemotherapy regimen given as part of a separate NCI breast cancer protocol. In such a case, prior approval of the principal investigator for that study should be obtained. It must be emphasized that no clinical or research endpoints of the chemotherapy protocol must be compromised by participation in this immune reconstitution protocol.

(2) In some cases, patients may receive non-experimental chemotherapy from their referring physicians. Patients may not be enrolled on this study if they are to receive chemotherapy as part of an experimental study performed outside of the NCI; patients who are receiving high-dose chemotherapy requiring stem cell support at other institutions are specifically excluded from participation in this study. The determination of whether non-experimental chemotherapy qualifies as dose intensive will be made by the principal investigator.

All stage II and III patients must represent a new diagnosis and must have received no prior chemotherapy.

Patients with metastatic disease can represent a new diagnosis as stage IV, or may have metastatic disease that represents a relapse after adjuvant therapy for any other stage of breast cancer. However, a prior of one year must have elapsed since the completion of adjuvant chemotherapy.

Patient must have a Hct of greater than or equal to 24%, a WBC count of greater than or equal to 3000 per mm(3), and platelets greater than or equal to 100,000 per mm(3) at the time of enrollment.

Patients must have no history of abnormal bleeding tendency or predisposition to infection.

Serum creatinine of less than 1.5 or Crcl of less than 60 cc per min. Higher values may be allowed if it is determined by the principal investigator that elevated values are due to tumor impairment of organ function.

AST and ALT less than 3 times the upper limits of normal. Higher values may be allowed if it is determined by the principal investigator that elevated values are due to tumor impairment of organ function.

In the presence of known pulmonary disease of symptoms, patients must have a pO2 greater than 65 and FEV1 and FVC greater than 65% of predicted (unless directly due to tumor involvement prior to therapy).

LVEF greater than or equal to 45% post-chemotherapy, as measured by MUGA or 2-D echocardiogram.

All patients must be free of a significant history or active symptomatology of coronary artery disease, congestive heart failure, neurologic disease, or chronic obstructive pulmonary disease.

Patients must have a Karnofsky performance score of greater than 70% (ECOG 0 or 1) and a life expectancy of at least three months.

Patients must be able to give informed consent.

POST-CHEMOTHERAPY ELIGIBILITY:

After completion of dose intensive chemotherapy, patients must continue to meet the eligibility criteria above. However, for patients who are to receive only autologous T cells (and no IL-2 therapy), cardiac ejection fraction will not represent a treatment eligibility criteria. In addition, patients must meet the criteria as outlined below.

To proceed with the protocol after completion of dose intensive chemotherapy, stage II and III patients must have no evidence of disease. Patients requiring adjuvant radiation therapy will receive this prior to proceeding with this protocol. Patients with metastatic disease must have demonstrated a least a partial response to chemotherapy (greater than 50% reduction in measurable disease).

To be eligible to proceed with T cell infusion and/or IL-2 administration after completion of chemotherapy, patients must have a Hb of greater than or equal to 9, an ANC greater than or equal to 1000, and a platelet count of greater than or equal to 75,000.

Patients must have recovered from any non-hematologic toxicities of dose-intensive chemotherapy and radiation therapy prior to receiving T cell infusions or IL-2.

All women will be tested for pregnancy at enrollment and prior to T cell transfer or IL-2 treatment; individuals must not be pregnant.

Patients must not be HIV positive or have Hepatitis B or C infection.

Patients must not have a chronic need to steroid or anti-coagulant therapy. However, for patients who are to receive only autologous T cells, steroid or anti-coagulant therapy will not be an exclusion criteria.

Patients must not present with any unusual medical or psychiatric risk.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51
Dates: Start 1995-07; Study Completion 2002-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Henderson IC, Hayes DF, Gelman R. Dose-response in the treatment of breast cancer: a critical review. J Clin Oncol. 1988 Sep;6(9):1501-15. doi: 10.1200/JCO.1988.6.9.1501. PMID 3047340
- [Background] Mackall CL, Fleisher TA, Brown MR, Magrath IT, Shad AT, Horowitz ME, Wexler LH, Adde MA, McClure LL, Gress RE. Lymphocyte depletion during treatment with intensive chemotherapy for cancer. Blood. 1994 Oct 1;84(7):2221-8. PMID 7919339
- [Background] Mackall CL, Fleisher TA, Brown MR, Andrich MP, Chen CC, Feuerstein IM, Horowitz ME, Magrath IT, Shad AT, Steinberg SM, et al. Age, thymopoiesis, and CD4+ T-lymphocyte regeneration after intensive chemotherapy. N Engl J Med. 1995 Jan 19;332(3):143-9. doi: 10.1056/NEJM199501193320303. PMID 7800006